CLINICAL TRIAL: NCT04672538
Title: Impact of Fontan Ventilation Strategy on Cardiac Output: An Invasive Physiologic Cross-over Study
Brief Title: Fontan Physiology Ventilation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Phillip S. Adams, DO, Assistant Professor of Anesthesiology, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20100012
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The trial will be a randomized crossover design.
Masking Description: Randomized cross over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low transition to High Vt protocol (Experimental): This arm of the study will begin with lower tidal volumes at higher respiratory rates for initial hemodynamic measurements. They will then be transitioned to the higher tidal volume at lower respiratory rate condition for repeat hemodynamic measurement.
  Interventions: Procedure: Low Vt protocol; Procedure: High Vt protocol
- High transition to Low Vt protocol (Experimental): This arm of the study will begin with higher tidal volumes at lower respiratory rates for initial hemodynamic measurements. They will then be transitioned to the lower tidal volume at higher respiratory rate condition for repeat hemodynamic measurement.
  Interventions: Procedure: Low Vt protocol; Procedure: High Vt protocol

INTERVENTIONS:
Procedure: Low Vt protocol — Low Vt protocol - tidal volumes (Vt) 6 ml/kg, respiratory rate required for end tidal carbon dioxide (EtCO2) of 36-38 mmHg, PEEP 5 centimeter of water (cm-H20) , I:E ratio 1:2
Procedure: High Vt protocol — High Vt protocol - tidal volumes (Vt) 10 ml/kg, respiratory rate required for EtCO2 of 36-38 mm Hg, PEEP 5 cmH2O, I:E ratio 1:3.

SUMMARY:
This study will investigate the different tidal volume (Vt) strategies during a cardiac catheterization procedure to determine whether or not low or high Vt have an impact on cardiac output.

Research question: While maintaining the same minute ventilation/PaCO2, does higher Vt (10 cc/kg)/lower rate vs. lower Vt (6 cc/kg)/higher rate (maintaining consistent PEEP) result in improved cardiac output?

DETAILED DESCRIPTION:
The trial will be a randomized crossover design. The study cohort will be randomized (50/50) to begin with either low Vt or high Vt ventilation. After achieving steady state, initial cardiac output measurements will be made using a measured oxygen consumption (VO2) and the Fick principle, per routine clinical protocol. Following baseline assessment of cardiac output and hemodynamics (which is standard of care for all catheterization procedures), participants will be transitioned to the alternative ventilation modality (high Vt or low Vt). After a 5-minute equilibration period, oxygen saturations and VO2 measurements will be re-acquired, to determine cardiac output and hemodynamics in this second state.

ELIGIBILITY:
Inclusion Criteria:

* Patients of UPMC Children's Hospital of Pittsburgh that have Fontan physiology (single heart ventricle) that are presenting as outpatients to undergo a cardiac catheterization with general endotracheal anesthesia for purpose of diagnosis or interventional cath.
* Parents and/or guardians willing to provide informed consent.

Exclusion Criteria:

* Those unwilling to give consent and those patients who do not have Fontan physiology.
* Any urgent/emergent catheterization procedure will be excluded.
* Any Fontan patient having a cardiac catheterization under monitored anesthesia care (as opposed to general endotracheal anesthesia) will not be eligible.
* Inability to undergo cardiac catheterization.
* Pregnant women will be excluded.
* < 6 weeks post-op from Fontan completion surgery
* Same hospitalization as Fontan completion surgery
* Intrinsic pulmonary disease which would be anticipated to impact study protocol / findings
* Fontan completion surgery performed at age > 7 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  The investigators will assess cardiac output using the Fink principle for each arm of randomization.

SECONDARY OUTCOMES:
Pulmonary blood flow | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  The investigators will compare blood flow in both arms.
Systemic blood pressure | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  The investigators will assess the vital sign in both intervention arms.
Pulmonary arterial pressure | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  The investigators will assess pressures in both intervention arms.
Pulmonary vascular resistance | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  Completed using pulmonary vascular resistance (PVR) equation from measurements obtained during the cardiac catheterization.
Systemic vascular resistance | Measurements will occur at the 5-minute equilibration period into the ventilation strategy.
  This will be calculated using appropriate equations using measurement obtained during catheterization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip S Adams, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shekerdemian LS, Bush A, Shore DF, Lincoln C, Redington AN. Cardiopulmonary interactions after Fontan operations: augmentation of cardiac output using negative pressure ventilation. Circulation. 1997 Dec 2;96(11):3934-42. doi: 10.1161/01.cir.96.11.3934. PMID 9403618